CLINICAL TRIAL: NCT05528549
Title: Blood Flow and Blood Pressure Investigation in Down Syndrome or Trisomy 21: FBI21
Brief Title: Blood Flow and Blood Pressure Investigation in Down Syndrome
Acronym: FBI21
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: American College of Sports Medicine (Other)
Responsible Party: Principal Investigator, Sara Rae Sherman, Graduate Student, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2022-0310
Record Dates: First submitted 2022-08-26; First posted 2022-09-06 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Down Syndrome
Keywords: Exercise; Blood Flow; Blood Pressure
MeSH Terms: conditions — Down Syndrome; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dynamic Exercise (Experimental): The investigators will look at leg blood flow during a seated leg-kicking test that is similar to biking. Leg blood flow will be measured in both the active and inactive legs. These measurements will be taken to examine how blood is directed (or controlled) during exercise.
  Interventions: Other: Exercise
- Static Exercise (Experimental): The investigators will look at blood pressure responses to a sustained leg kick. Blood pressure should increase during the sustained contraction for people without Down syndrome.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — The investigators are looking at how blood flow and blood pressure are regulated in individuals with Down syndrome, who have a reduced ability to do work. This study will compare individuals with Down syndrome to a control group without Down syndrome.

SUMMARY:
Down syndrome (DS) is a chromosomal condition that occurs in approximately 1 in 800 births worldwide, and causes impairments in physical function, including a reduced work capacity (as measured by VO2peak or aerobic capacity). Work capacity is important for activities of daily living, in order to live longer, healthier lives. Reduced work capacity stems in large part from autonomic dysfunction, which has been described in individuals with DS. Individuals with DS experience reduced sympathetic and parasympathetic control, which results in alterations in resting heart rate, blood pressure, and attenuated responses to sympathoexcitatory stimuli. Autonomic dysfunction may impair the ability to regulate blood flow and blood pressure to working muscles during exercise, which may cause a mismatch between oxygen supply and demand, further compromising the already reduced work capacity observed in individuals with DS. Utilization of a large muscle mass exercise, such as lower-limb dynamic exercise (similar to walking), requires a large shift in blood flow to match metabolic demand and allows the opportunity to evaluate blood flow regulation. Conversely, examination of the large changes in pressure in response to isometric exercise (i.e., a sustained contraction), allows for examination of the exercise pressor reflex as evoked by the isometric contraction. Thus, by comprehensively evaluating blood flow and blood pressure regulation, our work will further elucidate the mechanisms that underlay the reduced work capacity in individuals with DS. Improvement of overall work capacity for a population with reduced work capacity will guide future studies and exercise interventions aimed at helping to improve independence and quality of life, ultimately allowing individuals with DS to live longer, healthier lives.

Aim 1 (Dynamic Exercise): To examine the effects of an acute bout of dynamic leg kicking at both relative and absolute intensity workloads on femoral blood flow to both exercising and non-exercising muscle, in individuals with and without DS.

Aim 2 (Isometric Exercise): To examine the exercise pressor response to lower limb isometric exercise in individuals with and without DS.

DETAILED DESCRIPTION:
Specific Aims

Down Syndrome (DS) is the most prevalent genetic form of intellectual disability, and individuals with DS have low work capacity. Reduced work capacity limits gross motor function, and thus, reduces independence, full participation, and ultimately quality of life (QOL). Low work capacity is associated with central autonomic dysfunction in persons with DS, which limits maximal heart rates ~30 beats below expected values. However, during exercise, the autonomic nervous system also balances peripheral blood flow delivery and blood pressure regulation, through the redistribution of blood to active skeletal muscle. Blood flow redistribution occurs primarily through sympathetically-mediated changes in vasomotor tone by stimulation of mechanically and metabolically sensitive afferent fibers in the skeletal muscle, which results in changes in pressure to maintain adequate flow. It is unknown whether the observed central autonomic dysfunction in individuals with DS also alters peripheral blood flow regulation or the blood pressure response to lower limb exercise, which is critical to improving work capacity and ultimately participation and QOL.

Blood flow redistribution occurs in an intensity-dependent manner regulated through changes in pressure, away from inactive tissue towards exercising or active muscle through vasoconstrictive mechanisms. Data from our lab using a mild sympathetic stimulus, namely lower body negative pressure, suggests individuals with DS have reduced vasoconstrictive control. Reduced ability to vasoconstrict inactive tissue during exercise may inhibit appropriate distribution of blood flow to active muscle, which may be particularly limiting during large muscle exercise, thereby limiting work capacity. In addition to reduced vasoconstrictive control, blood flow during exercise is driven by sympathetically-mediated increases in blood pressure from muscular contraction activating the mechano- and metaboreflexes, termed the exercise pressor reflex. Individuals with DS have a blunted blood pressure response to sympathoexcitatory challenges, such as isometric handgrip exercise, suggesting impairments in blood pressure regulation. Taken together, our previous work (i.e., preliminary data) suggests that the redistribution of blood flow and blood pressure regulation may be impaired during stimuli involving small muscle mass for individuals with DS. However, blood flow and blood pressure regulation have not been examined using large muscle exercise (e.g., lower limb exercise) in DS, which may be a more impactful and limiting factor for individuals with DS in regards to work capacity.

Active, lower limb exercise requires greater peripheral blood flow regulation to ensure a match between oxygen demand and supply, which is critical to improving blood pressure regulation and thus, work capacity. The aim of this study is to comprehensively evaluate blood flow redistribution by examining blood flow to active and non-active legs during dynamic (rhythmic muscular activity) lower limb exercise with increasing exercise intensity. In contrast, isometric (contraction of muscles without movement in surrounding joints) lower limb exercise will allow for investigation of blood pressure regulation in individuals with DS through activation of the exercise pressor reflex. More specifically, the metaboreflex can be assessed with post-exercise ischemia that traps metabolites in a regional area, wherein blood pressure and sympathetic activity remain elevated, independent of cardiac output. Interestingly, neither blood flow redistribution nor the exercise pressor response to large muscle exercise have been previously explored in individuals with DS. Investigation of these mechanisms will help elucidate the mechanisms of low work capacity, ultimately leading to improved health outcomes, participation, and QOL for individuals with DS.

The overall aim of this study is to comprehensively evaluate blood flow regulation, including the pressor reflex, in two research aims: Aim 1 (Dynamic Exercise): To examine the effects of lower limb dynamic exercise on femoral blood flow in both exercising and non-exercising legs in individuals with and without DS. The investigators hypothesize individuals with DS will have: a) attenuated femoral blood flow to the active leg at all intensity workloads of dynamic exercise and b) a lack of blood flow control as demonstrated by a lack of vasoconstriction in the non-exercising leg compared to individuals without DS. Aim 2 (Isometric Exercise): To examine the effects of lower limb isometric exercise on the exercise pressor response in individuals with and without DS. The investigators hypothesize the individuals with DS will exhibit an attenuated blood pressure response, demonstrating dysfunction of the exercise pressor reflex following isometric single-leg extension.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 yrs old and apparently healthy individuals
* Mild to moderate intellectual disability for individuals with DS
* Corrected congenital heart disease for individuals with DS
* Euthyroid or on stable thyroid medication for at least 6 months
* Free from cardiovascular, pulmonary, inflammatory, or metabolic disease
* BMI <40kg/m2

Exclusion Criteria:

* Hypertension (resting systolic blood pressure [SBP] ≥140 and/or diastolic blood pressure [DBP] ≥90 mmHg) this includes those on medications to treat hypertension
* Hypotension (resting blood pressure [BP] of <90/60 mmHg)
* Cancer in the last 6 months
* Any heart-rate-altering medications or any other medication that may modify metabolic responses
* Anti-inflammatory medication for 7 days prior to testing
* Self-reported diabetes or use of glucose lowering medication
* Tobacco products, including vaping, or marijuana use
* Premenopausal women who use non-oral contraceptives
* Non-English speakers
* Currently pregnant
* Inability to perform leg extension exercises or any orthopedic limitations that would prohibit seated, stationary leg kicking

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-04-26 (Actual); Study Completion 2023-04-26 (Actual)

PRIMARY OUTCOMES:
Blood Flow | During study visit 1, lower limb blood flow will be measured as a change from baseline to blood flow during leg contraction. It will also be measured as a change from baseline to post leg contraction blood flow.
  The investigators will use a Doppler ultrasound machine to assess lower limb blood flow during repeated leg contractions.
Blood Pressure | During study visit 2, blood pressure will be measured as a change from baseline blood pressure to leg contraction blood pressure. It will also be measured as a change in baseline blood pressure to post leg contraction blood flow.
  The investigators will continuously measure blood pressure during a static leg contraction.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Motl, Ph.D., Study Chair — University of Illinois at Chicago; Tracy Baynard, Ph.D., Study Chair — University of Massachusetts at Boston
Locations (1):
- Disability, Health & Social Policy Building; Integrative Physiology Lab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sherman SR, Jackson RE, Hibner BA, Lima NS, Cloud RM, Fernhall B, Baynard T. Blunted exercise hyperemic response to lower limb exercise in individuals with Down syndrome. Am J Physiol Heart Circ Physiol. 2025 Aug 1;329(2):H374-H387. doi: 10.1152/ajpheart.00080.2025. Epub 2025 Jun 30. PMID 40588365
- [Derived] Sherman SR, Jackson R, Lima NS, Hibner BA, Fernhall BO, Baynard T. Blunted Exercise Pressor Response to Isometric Knee Extension and Post-Exercise Ischemia in Individuals with Down Syndrome. Med Sci Sports Exerc. 2025 Apr 1;57(4):876-883. doi: 10.1249/MSS.0000000000003619. Epub 2024 Dec 3. PMID 39625363